CLINICAL TRIAL: NCT06947694
Title: A Prospective, Multicenter, Umbrella Design Clinical Study on the Abscopal Effect Induced by Different Radioimmunotherapy Combination Patterns in the Treatment of Non-Small Cell Lung Cancer With Multiple Metastases
Brief Title: A Study on Exploring the Abscopal Effect Induced by Different Radioimmunotherapy Combination Patterns in the Treatment of Non-Small Cell Lung Cancer With Multiple Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, prof, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-024
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV Without EGFR/ALK Mutation
MeSH Terms: interventions — Drug Therapy; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group A (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group B (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group C (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group D (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group E (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group F (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors
- Group G (Experimental)
  Interventions: Drug: chemotherapy + PD-1 inhibitors

INTERVENTIONS:
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8Gy * 3-10 fractions) for pulmonary lesions, lymph node lesions and visceral lesions in combination with the PD-1 inhibitors . During the follow-up, the PD-1 inhibitors will be maintained until the disease progresses or the toxicity is intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group A
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8 Gy × 3-10 fractions) for pulmonary lesions, lymph node lesions and other lesions in combination with the PD-1 inhibitors. During the follow-up, the PD-1 inhibitors will be continued until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group B
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8Gy × 3-10 fractions) for pulmonary lesions, lymph node lesions and bone metastatic lesions in combination with the PD-1 inhibitors . During the follow-up, the PD-1 inhibitors will be continued until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group C
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8 Gy × 3-10 fractions) for pulmonary lesions, visceral lesions and other lesions in combination with the PD-1 inhibitors. During the follow-up, the PD-1 inhibitors will be maintained until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group D
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8 Gy × 3-10 fractions) for pulmonary lesions, visceral lesions and bone metastatic lesions in combination with the PD-1 inhibitors. During the follow-up, the PD-1 inhibitors will be continued until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group E
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8 Gy × 3-10 fractions) for lymph node lesions, visceral lesions and other lesions in combination with the PD-1 inhibitors. During the follow-up, the PD-1 inhibitors will be continued until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group F
Drug: chemotherapy + PD-1 inhibitors — The patient receives 4 cycles of treatment with "chemotherapy + PD-1 inhibitors". If there is no disease progression, the patient will receive radiotherapy (radiation dose: 5-8 Gy × 3-10 fractions) for lymph node lesions, visceral lesions and other lesions in combination with the PD-1 inhibitors. During the follow-up, the PD-1 inhibitors will be continued until the disease progresses or the toxicity becomes intolerable. The maximum duration of immunotherapy shall not exceed 2 years.
  Other Names: Radiotherapy
  Arms: Group G

SUMMARY:
It is planned to carry out a multicenter umbrella study to find the optimal organ combination and the best radioimmunotherapy combination pattern, so as to improve the survival of NSCLC patients with multiple metastases. At the same time, by using multimodal omics data, machine learning will be employed to construct a prediction model for the abscopal effect, and explore the immunoregulation of organ-specific radiotherapy and biomarkers of the abscopal effect. The main objective is to find the optimal organ combination and the best radioimmunotherapy combination pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet all of the following inclusion criteria to be enrolled in this study:

  1. Non-small cell lung cancer diagnosed initially through pathological histology.
  2. There are 3-6 metastatic lesions.
  3. No brain metastasis or the lesions are stable.
  4. Negative for driver genes (including EGFR, ALK, ROS, BRAF, MET, RET genes. Note: The above English terms are all gene names).
  5. ECOG (Eastern Cooperative Oncology Group) score: 0-1 point, with an expected, survival period of more than 3 months.
  6. Aged between 18 and 75 years old.
  7. Evaluated by PET-CT (including FDG and FMISO, not mandatory).
  8. No contraindications for immunotherapy and radiotherapy.
  9. The informed consent form has been signed.

Exclusion Criteria:

* Patients with any of the following criteria are not eligible for enrollment in this study:

  1. Those with severe dysfunction of vital organs (heart, liver, kidney).
  2. Those accompanied by other malignant tumors.
  3. Those with uncontrolled heart diseases or having experienced a myocardial infarction within the past six months.
  4. Those with a history of mental illness.
  5. And other situations in which the researchers deem it inappropriate for the subjects to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The remission rate of abscopal lesions | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
  The remission rate of abscopal lesions. Immunotherapy is administered within less than 1 week after the start of radiotherapy. The time point for determining the abscopal effect is set as ≤ 4 cycles of immunotherapy. The assessment is carried out in accordance with the RECIST 1.1 (Appendix 1) and iPERCIST criteria.

SECONDARY OUTCOMES:
PFS | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
OS | up to 5 years
ORR | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
DOR | From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
irAE | From date of consent informed until 60 days after the last investigational product administration. Up to 2 approximately years
  Adverse reactions related to immunotherapy
QoF | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Sun, MD, Principal Investigator — the second affiliated hospital of Army medical university, Chongqing, Chongqing 40037 Recruiting
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No